CLINICAL TRIAL: NCT06445491
Title: Influence of Test Order of Isokinetic Torque, Y-Balance/Firefighter-Specific Functional-Balance, and Forward-Step-Down on Test Performance: Identifying Optimal Sequences
Brief Title: Effect of Sequencing on Outcome Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00002716
Record Dates: First submitted 2024-05-22; First posted 2024-06-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Muscle Weakness
Keywords: strength; dynamic balance; movement quality; injury prevention
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: All participants will receive all 6 iterations of testing order, but the order of test sequences will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control trial (Active Comparator): Testing order: (1) forward step down test, (2) firefighter specific functional balance test & y-balance test, (3) hip isokinetic strength & knee isokinetic strength
  Interventions: Other: Control order
- sequenced trials (Experimental): Participants will perform the following variations on testing order over 6 separate sessions: 1-2-3, 1-3-2, 2-1-3, 2-3-1, 3-1-2, and 3-2-1
  Interventions: Other: Randomized sequence

INTERVENTIONS:
Other: Control order — Participants will perform an initial baseline of tests, order of 1- 2- 3
  Arms: control trial
Other: Randomized sequence — the testing order will be randomized for follow up testing.
  Arms: sequenced trials

SUMMARY:
This pilot study will examine the effect of testing order on test outcomes for measures of strength, dynamic balance, and movement quality. Each participant will perform a baseline test, then will perform the 6 iterations of the testing sequence.

DETAILED DESCRIPTION:
This study employs a Repeated Measures Design, with each participant tested multiple times in combinations of 1) the Isokinetic Torque Test, 2) the Y-Balance Test/Firefighter-Specific Functional-Balance Test, and 3) the Forward-Step-Down Test. The investigators will conduct a total of seven testing sessions, including a control session (informed consent, familiarization with outcome measures, and control data collection) and the following six different patterns: 1-2-3, 1-3-2, 2-1-3, 2-3-1, 3-1-2, and 3-2-1. The order of the sessions will be randomized and counterbalanced to prevent bias effects. The control session will be performed in the following order: (1) Forward-Step-Down Test, (2a) Firefighter Specific Functional Balance Test, (2b) Y-balance test, (3) isokinetic tests (hip then knee).

Participants will be asked to avoid exercise or vigorous physical activity for the 24 hours prior to any testing session to minimize the effects of non-test-related fatigue on the study outcomes. Pre and post-test fatigue will be measured with the Rating of Fatigue (ROF) Scale. Pre-and post-test exertion will be measured with the Borg Rating of Perceived Exertion (RPE) Scale (attached). Heartrate will be measured and recorded at each scale rating point.

Upon arrival for the control session, participants will have their height measured using a stadiometer and their weight recorded. This will be followed by the performance of the initial 1-2-3 pattern. The time needed for the participant to perform each test will be recorded and subsequent performances of that test will be carried out in this time frame.

For visits two through seven, participants will be weighed again upon arrival and perform one of the six patterns. Sessions two to seven will be separated by at least one day to minimize the influence of fatigue. Each session will include isokinetic torque measurements of the hip abductors and adductors, knee flexors and extensors, the Y-Balance Test, the Firefighter-Specific Functional-Balance Test, and the Forward-Step-Down Test. The dominant leg will be used for unilateral tests, as determined by the leg used to kick a ball. The order of outcome measures will be randomized for each participant to minimize the effects of fatigue and recovery.

Five minutes of warm-up on a stationary bike or walking will be performed to start each exercise session. Five minutes of rest and instruction will be provided between each outcome measure. Five minutes of rest will be given between isokinetic tests (hip abduction to adduction) to allow for machine set-up and instructions. One minute of rest will be given between each isokinetic speed, with three speeds tested for the hip (30°, 60°, and 120° per second) and knee (60°, 180°, and 300° per second) muscles.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult by Physical Activity Readiness Questionnaire+ screening process

Exclusion Criteria:

* lower extremity or spine injury in past 6 months
* vestibular disorder
* known pregnancy
* inability to complete data collection

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Forward-Step-Down Test | This outcome will be assessed at each visit throughout the study, an average of 6 weeks.
  a step-down task that is performed off a 20 cm box. Five repetitions are performed to give one score (minimum score 0, maximum score 6). A higher score is worse.
Firefighter Specific Functional Balance Test | This outcome will be assessed at each visit throughout the study, an average of 6 weeks.
  A dynamic balance test performed by stepping down from a 15cm box, walking across a low beam (4cm high), and stepping up onto a 10cm box, turning around, and returning to the original box. 8 Trials are performed. In 4 trials, a bar is placed at 75% of the participant's height for them to negotiate while on the beam. A faster time with fewer errors is better.
Y-Balance Test | This outcome will be assessed at each visit throughout the study, an average of 6 weeks.
  A dynamic balance test that is performed on the dominant leg, reaching in the anterior, posteromedial, and posterolateral directions. The length of reach is standardized to participants' leg length. A higher score is better.
Knee Extensor Isokinetic Test | This outcome will be assessed at each visit throughout the study, an average of 6 weeks.
  Knee extensor isokinetic strength will be tested at 60°, 180°, and 300° per second from the seated position with 5, 10, and 10 concentric contractions for each speed. A higher reading of strength is better.
Hip Abductor Isokinetic Test | This outcome will be assessed at each visit throughout the study, an average of 6 weeks.
  Hip abductor strength will be tested at 30°, 60°, and 120° per second from the standing position. A higher reading of strength is better.

SECONDARY OUTCOMES:
Rating of Fatigue | This outcome will be assessed at each visit throughout the study, an average of 6 weeks.
  A score from 0-10 will be provided before and after each test category (strength, balance, movement quality). A higher score indicated more fatigue.
Rating of Perceived Exertion | This outcome will be assessed at each visit throughout the study, an average of 6 weeks.
  A score from 6-20 will be provided before and after each test category (strength, balance, movement quality). A higher score indicated more perceived exertion.
Heartrate | This outcome will be assessed at each visit throughout the study, an average of 6 weeks.
  heartrate will be recorded as a measure of physiological effort and for participant safety.

CONTACTS AND LOCATIONS:
Overall Officials: Erin McCallister, DPT, Principal Investigator — LSUHSC-Shreveport
Locations (1):
- LSUHSC-Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gagge AP, Stolwijk JA, Hardy JD. Comfort and thermal sensations and associated physiological responses at various ambient temperatures. Environ Res. 1967 Jun;1(1):1-20. doi: 10.1016/0013-9351(67)90002-3. No abstract available. PMID 5614624
- [Background] Games KE, Winkelmann ZK, McGinnis KD, McAdam JS, Pascoe DD, Sefton JM. Functional Performance of Firefighters After Exposure to Environmental Conditions and Exercise. J Athl Train. 2020 Jan;55(1):71-79. doi: 10.4085/1062-6050-75-18. Epub 2019 Dec 26. PMID 31876454
- [Background] Hewett TE, Ford KR, Hoogenboom BJ, Myer GD. Understanding and preventing acl injuries: current biomechanical and epidemiologic considerations - update 2010. N Am J Sports Phys Ther. 2010 Dec;5(4):234-51. PMID 21655382
- [Background] Lopes TJA, Simic M, Myer GD, Ford KR, Hewett TE, Pappas E. The Effects of Injury Prevention Programs on the Biomechanics of Landing Tasks: A Systematic Review With Meta-analysis. Am J Sports Med. 2018 May;46(6):1492-1499. doi: 10.1177/0363546517716930. Epub 2017 Jul 31. PMID 28759729
- [Background] Nascimento LR, Teixeira-Salmela LF, Souza RB, Resende RA. Hip and Knee Strengthening Is More Effective Than Knee Strengthening Alone for Reducing Pain and Improving Activity in Individuals With Patellofemoral Pain: A Systematic Review With Meta-analysis. J Orthop Sports Phys Ther. 2018 Jan;48(1):19-31. doi: 10.2519/jospt.2018.7365. Epub 2017 Oct 15. PMID 29034800
- [Background] Park KM, Cynn HS, Choung SD. Musculoskeletal predictors of movement quality for the forward step-down test in asymptomatic women. J Orthop Sports Phys Ther. 2013;43(7):504-10. doi: 10.2519/jospt.2013.4073. Epub 2013 Jun 11. PMID 23756380
- [Background] McCallister, E., & Flowers, D. W. (2020). Can the Forward-Step-Down Test Be Used Reliably in the Clinical Setting to Assess Movement Changes Resulting from Maximal Exertion? A Pilot Study. Internet Journal of Allied Health Sciences and Practice, 18(4).
- [Background] Powers CM. The influence of abnormal hip mechanics on knee injury: a biomechanical perspective. J Orthop Sports Phys Ther. 2010 Feb;40(2):42-51. doi: 10.2519/jospt.2010.3337. PMID 20118526
- [Background] van Melick N, Meddeler BM, Hoogeboom TJ, Nijhuis-van der Sanden MWG, van Cingel REH. How to determine leg dominance: The agreement between self-reported and observed performance in healthy adults. PLoS One. 2017 Dec 29;12(12):e0189876. doi: 10.1371/journal.pone.0189876. eCollection 2017. PMID 29287067
- [Background] Brent JL, Myer GD, Ford KR, Paterno MV, Hewett TE. The effect of sex and age on isokinetic hip-abduction torques. J Sport Rehabil. 2013 Feb;22(1):41-6. doi: 10.1123/jsr.22.1.41. Epub 2012 Jun 18. PMID 22715125
- [Background] Claiborne TL, Timmons MK, Pincivero DM. Test-retest reliability of cardinal plane isokinetic hip torque and EMG. J Electromyogr Kinesiol. 2009 Oct;19(5):e345-52. doi: 10.1016/j.jelekin.2008.07.005. Epub 2008 Oct 8. PMID 18845450
- [Background] Gokeler A, Welling W, Zaffagnini S, Seil R, Padua D. Development of a test battery to enhance safe return to sports after anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2017 Jan;25(1):192-199. doi: 10.1007/s00167-016-4246-3. Epub 2016 Jul 16. PMID 27423208